CLINICAL TRIAL: NCT06666894
Title: Intermittent Fasting Versus Dietary Approach to Stop Hypertension on Metabolic Risk Profile in Nonalcoholic Fatty Liver Patients
Brief Title: Intermittent Fasting Versus Diet to Stop Hypertension on Metabolic Risk Profile in Nonalcoholic Fatty Liver Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Khattab Omer, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aya-005258
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Fasting, Intermittent; Diet; Hypertension; Metabolic Syndrome; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Intermittent Fasting; Hypertension; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting group (Experimental): intermittent fasting time-restricted feeding (TRF) subjects consumed 100 % of their energy needs in an 8 hours period of time each day, with their caloric intake divided into three meals consumed at 1 p.m., 4 p.m., and 8 p.m. schedule (8-hr daily eating period, The remaining 16 hours per 24-hour period made up the fasting period)
  Interventions: Other: Intermittent fasting
- Diet group (Active Comparator): the dietary approach to stop hypertension (DASH) subjects consumed 100 % of their energy needs divided into three meals consumed at 8 a.m., 1 p.m., and 8 p.m. (12-hr eating period).
  Interventions: Other: Dietary approach to stop hypertension (DASH)

INTERVENTIONS:
Other: Intermittent fasting — subjects consumed 100 % of their energy needs in an 8-h period of time each day, with their caloric intake divided into three meals consumed at 1 p.m., 4 p.m., and 8 p.m. The remaining 16 h per 24-h period made up the fasting period. Subjects in the ND group consumed 100 % of their energy needs divided into three meals consumed at 8 a.m., 1 p.m., and 8 p.m. all patients will be subjected to 30 minutes mild aerobic exercise on treadmill.
  Arms: Intermittent fasting group
Other: Dietary approach to stop hypertension (DASH) — The USDA's 2015-2020 Dietary Guidelines for Americans recommend a healthy eating pattern, including a variety of vegetables, fruits, whole grains, fat-free dairy, protein, and oils. Limit saturated fats, trans fats, added sugars, and sodium to less than 10% daily calories, 10% saturated fat daily calories, and 2,300 mg sodium per day.
  Arms: Diet group

SUMMARY:
This study was conducted to compare between the effect of intermittent fasting and diatery approach to stop hypertension on metabolic risk profile in nonalcoholic fatty liver patients.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver is a liver disease linked to obesity, insulin resistance, type 2 diabetes, hypertension, hyperlipidemia, and metabolic syndrome. The subtype, non-alcoholic steatohepatitis, can lead to liver fibrosis, cirrhosis, hepatocellular carcinoma, and liver transplantation. The prevalence of Non-alcoholic fatty liver disease is increasing at the same rate as obesity, with the global prevalence estimated at 25%. By 2020, the burden of Non-alcoholic fatty liver is expected to exceed that of communicable disease in most regions.

ELIGIBILITY:
Inclusion Criteria:

* Non-alcoholic fatty liver patients diagnosed by radiological ultrasound
* BMI >30
* All patients are sedentary lifestyle with little or no exercise.
* High lipid profile (total cholesterol > 200, LDL > 130, TAGs > 150) patients by laboratory investigation.
* High fasting insulin level > 20mlU/mL & high fasting Glucose level >100, HbA1c > 5.7 & high HOMA- IR > 2.5 patients by Laboratory investigation.
* High inflammatory markers (IL6) patients.
* Age ranged from 30 to 40 years old.

Exclusion Criteria:

* Alcoholic fatty liver patients.
* Cirrhosis patients.
* Diabetes patients.
* Cognitive impaired patients.
* History of epilepsy patients.
* Cardiac pacemaker patients.
* Anemic patients
* pregnancy

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
assessment of Non-alcoholic fatty liver using ultrasonography | at baseline at after two months
  usage of diagnostic ultrasound to diagnose patients with non-alcoholic fatty liver disease

SECONDARY OUTCOMES:
assessment of change of lab profile using laboratory investigations | at baseline at after two months
  The study focuses on lipid profiles, glucose and insulin profiles, IL-6, and C- reactive protein. Blood samples are collected from the antecubital vein at baseline and after 8 weeks, and analyzed using the same reagent lot. Fasting total cholesterol, HDL-C, LDL-C, and triglycerides are measured using an enzymatic colorimetric method. LDL-C fraction is calculated using Friedewald's formula. Laboratory investigation before and after the study is conducted.
assessment of change of body mass index | at baseline at after two months
  Anthropometric baseline characteristics of subjects by In Body 170 Pre & post the study being performed (BMI)
assessment of macronutrients distribution | at baseline at after two months
  • Dietary assessment for macronutrients distribution by dietary 24-hour recall Highlighted among dietary assessment methods of the current diet for their interest & validity. It is a prospective, open ended survey method collecting data about the foods & beverages consumed over a previously specified period of time.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Giza, Egypt